CLINICAL TRIAL: NCT05624125
Title: BEETroot Juice to Reverse Functional Impairment in PAD: The BEET PAD Trial
Brief Title: BEETroot Juice to Reverse Functional Impairment in PAD
Acronym: BEET PAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Virginia (Other); University of Chicago (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Mary McDermott, Jeremiah Stamler Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00217101; R01AG073257 (NIH)
Record Dates: First submitted 2022-11-13; First posted 2022-11-21 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Peripheral Artery Disease
Keywords: beetroot juice, mobility, intermittent claudication, peripheral artery disease
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot juice (Active Comparator): The beetroot juice intervention comes in a single 70 ml drink and is manufactured by James White Drinks. Each drink contains beetroot juice and 2% lemon juice, made from concentrates. Each serving of 70 mL of beetroot juice contains 400 mgs (6.45 millimoles) of nitrate and will be taken twice daily for a total daily dose of 800 mgs (12.90 millimoles) of nitrate.
  Interventions: Other: Beetroot juice
- Placebo (Placebo Comparator): The placebo comes in a single 70 ml drink and is manufactured by James White Drinks. The placebo contains beetroot juice and 2% lemon juice, made from concentrates, and is filtered to remove nitrate.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Beetroot juice — Two 70 ml beetroot juice drinks daily for 4 months.
  Arms: Beetroot juice
Other: Placebo — Two 70 ml placebo drinks daily for 4 months.
  Arms: Placebo

SUMMARY:
The BEET PAD Trial is a multi-centered double-blind randomized clinical trial designed to determine whether beetroot juice, compared to placebo, improves six-minute walk distance at four month follow-up in people with lower extremity peripheral artery disease (PAD). Investigators hypothesize that by simultaneously increasing lower extremity perfusion, gastrocnemius muscle mitochondrial activity, and myofiber health and regeneration, beetroot juice will significantly improve walking performance in people with PAD. The primary aim is to determine whether beetroot juice significantly improves six-minute walk distance at 4-month follow-up in people with PAD, compared to placebo. Preliminary evidence suggests that beetroot juice has both acute and chronic effects on walking performance in PAD. The primary outcome will measure the combined acute and chronic effect of beetroot juice (i.e. the maximal effect) on change in 6-minute walk at 4-month follow-up. In secondary aims, investigators will distinguish between acute and chronic effects of beetroot juice on six-minute walk and delineate biologic pathways by which beetroot juice improves walking performance in PAD, by measuring change in gastrocnemius muscle perfusion (MRI arterial spin labeling) and gastrocnemius muscle health. The trial will assess the durability of beetroot juice effects on six-minute walk. Nitrate in beetroot juice is metabolized to nitrite and subsequently to NO, attaining peak nitrite levels 2.5 hours after ingestion. The trial will determine whether a higher peak or a greater increase in plasma nitrite at 2.5 hours after beetroot juice consumption at baseline has a greater effect on six-minute walk at 4-month follow-up, compared to a lower peak or a smaller increase, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 and older
2. Presence of peripheral artery disease, defined as:

   1. An ankle brachial index (ABI) <= 0.90 at baseline
   2. Vascular lab evidence of PAD (such as a toe brachial pressure <= 0.70 or an ankle brachial index <=0.90), or angiographic evidence of PAD defined as at least 70% stenosis of an artery supplying the lower extremities.
   3. An ABI of >0.90 and <=1.00 who experience a 20% or greater drop in ABI in either leg after the heel-rise test.

Exclusion Criteria:

1. Above- or below-knee amputation
2. Critical limb ischemia defined as an ABI <0.40 with symptoms of rest pain
3. Wheelchair confinement or requiring a walker to ambulate
4. Walking is limited by a symptom other than PAD
5. Current foot ulcer on bottom of foot
6. Failure to successfully complete the study run-in
7. Planned major surgery, coronary or leg revascularization during the next five months
8. Major surgery, coronary or leg revascularization or major cardiovascular event in the previous three months
9. Major medical illness including lung disease requiring oxygen, Parkinson's disease, a life-threatening illness with life expectancy less than six months, or cancer requiring treatment in the previous two years. [NOTE: potential participants may still qualify if they have had treatment for an early stage cancer in the past two years and the prognosis is excellent. Participants who require oxygen only at night may still qualify.]
10. Mini-Mental Status Examination (MMSE) score < 23
11. Allergy to beetroot juice
12. Currently consuming beetroot juice, oral nitrate or nitrite, or a beetroot supplement and/or unwilling to avoid beetroot juice during the study. Participants will be asked to discontinue these items for 30 days before baseline testing and throughout the clinical trial. If the potential participant is unwilling to refrain from taking these items, they will not be eligible for the clinical trial.
13. Currently consuming one cup or more of beets daily. Participants will be asked to discontinue beet ingestion of one cup or more of beets for 30 days before baseline testing and throughout the clinical trial. If the potential participant is unwilling to refrain from daily beet consumption of one cup or more for 30 days before the trial and during the trial, they will not be eligible for the clinical trial.
14. Non-English speaking
15. Participation in or completion of a clinical trial in the previous three months. [NOTE: after completing a stem cell or gene therapy intervention, participants will become eligible after the final study follow-up visit of the stem cell or gene therapy study so long as at least six months have passed since the final intervention administration. After completing a supplement or drug therapy (other than stem cell or gene therapy), participants will be eligible after the final study follow-up visit as long as at least three months have passed since the final intervention of the trial.]
16. Visual impairment that limits walking ability.
17. Six-minute walk distance of <500 feet or >1600 feet. Investigator discretion will be used to decide whether participants who walk greater than 1600 feet are eligible.
18. Baseline blood pressure <100/45.
19. Participation in a supervised treadmill exercise program in previous three months.
20. Using an antibacterial mouthwash (such as Cepacol) or a mouthwash containing chlorhexidine and unwilling to discontinue.
21. In addition to the above criteria, investigator discretion will be used to determine if the trial is unsafe or not a good fit for the potential participant.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Four-month change in six-minute walk distance | Baseline to four-month follow-up
  Change in six-minute walk distance at four-month follow-up will be compared between those randomized to beetroot juice vs. those randomized to placebo

SECONDARY OUTCOMES:
2.5 hour change in six-minute walk distance (acute effect) | Baseline 2.5 hour follow-up
  Change in six-minute walk distance 2.5 hours after drinking the first study beverage (acute effect) will be compared between those randomized to beetroot juice vs. those randomized to placebo
Four-month + 24 hour change in six-minute walk distance (chronic effect) | Baseline to four-month + 24 hour follow-up
  Change in six-minute walk distance at four-month follow-up, 24 hours after drinking study beverage (chronic effect) will be compared between those randomized to beetroot juice vs. those randomized to placebo
Four-month change in calf muscle perfusion | Baseline to four-month follow-up
  Change in calf muscle perfusion will be compared between those randomized to beetroot juice vs. those randomized to placebo
Four-month change in Walking Impairment Questionnaire (WIQ) distance score | Baseline to four-month follow-up
  Change in WIQ distance score will be compared between those randomized to beetroot juice vs. those randomized to placebo
Four-month change in six-minute walk distance among participants randomized to beetroot juice | 2.5 hour to four-month follow-up
  Among those randomized to beetroot juice, investigators will determine whether those who attain a higher immediate peak or a greater increase in plasma nitrate levels at 2.5 hours after the first dose of beetroot juice at baseline will have a greater six-minute walk improvement at 4-month follow-up, compared to those with a lower peak or a smaller increase in nitrite, respectively

OTHER OUTCOMES:
Durability of effect on six-minute walk distance | 14 days after the end of the assigned study drink (intervention or placebo)
  Change in six-minute walk distance at 14 days after the final drink that the participant was randomized to will be compared between those randomized to beetroot juice vs. those randomized to placebo
Four-month change in Walking Impairment Questionnaire (WIQ) speed and stair climbing scores | Baseline to four-month follow-up
  Change in WIQ speed and stair climbing scores at four-month follow-up will be compared between those randomized to beetroot juice vs. those randomized to placebo
Four-month change in Short-Form 36 Physical Function questionnaire score | Baseline to four-month follow-up
  Change in Short-Form 36 Physical Function questionnaire score at four-month follow-up will be compared between those randomized to beetroot juice vs. those randomized to placebo
Four-month change in short physical performance battery (SPPB) score | Baseline to four-month follow-up
  Change in SPPB score at four-month follow-up will be compared between those randomized to beetroot juice vs. those randomized to placebo
Four-month change in nitrate and nitrite abundance in muscle | Baseline to four-month follow-up
  Change in nitrate and nitrate abundance in muscle in participants who undergo gastrocnemius (calf) muscle biopsy will be compared between those randomized to beetroot juice vs. those randomized to placebo
Four-month change in mitochondrial oxygen consumption | Baseline to four-month follow-up
  Change in mitochondrial oxygen consumption in participants who undergo gastrocnemius (calf) muscle biopsy will be compared between those randomized to beetroot juice vs. those randomized to placebo

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No